CLINICAL TRIAL: NCT01745809
Title: An Exploratory Study to Obtain Functional and Transcriptional/Translational Profiling of Cells From Bronchial Lavages and Brushings in Severe Asthmatics and Healthy Control Subjects
Brief Title: Bronchoscopy Study for Severe Asthma
Status: Withdrawn | Type: Observational
Why Stopped: Contractual issues
Sponsor: University of Pennsylvania (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 814383
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2011-10

CONDITIONS: Severe Persistent Asthma
MeSH Terms: interventions — Bronchoscopy; Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Severe Asthmatics: Subjects with a pre-existing physician diagnosis of asthma with reversible airflow obstruction of at least 12%.
  Interventions: Procedure: Bronchoscopy
- Healthy non-smokers: Subjects will be never smokers or former smokers for the past year and less than 10 pack years lifetime with no history of asthma or any other lung disease.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Subjects will have a screening visit and, if they qualify to take part in the study, they will undergo a single bronchoscopy procedure. During the bronchoscopy, bronchoalveolar lavage (BAL) and bronchial brushings will be performed on each subject.
  Other Names: Fiberoptic Bronchoscopy; Bronchoalveolar Lavage

SUMMARY:
The purpose of this research study is to collect lung tissue and fluid from two groups of people: those who have severe asthma, and those who do not. These samples will then be tested in a laboratory to identify differences in the lung tissue cells and fluids that may exist between these two groups of people.

ELIGIBILITY:
Inclusion Criteria:

* Asthma Subject Inclusion Criteria

  1. Subject is an adult male or female between 18 and 65 years of age inclusive.
  2. Subject must have a pre-history of a physician's diagnosis of severe asthma (according to GINA classification) with some reversible airway obstruction (shown by peak flow or FEV1 in the last 12 months with a change of 12% in the absolute FEV1 measurement) and an exclusion of other significant pulmonary diseases (i.e., cystic fibrosis, tuberculosis, Interstitial Lung Disease and bronchopulmonary dysplasia)
  3. Subject has a positive methacholine test (PC20 < 16). This test sometimes cannot be performed in severe asthmatics because of low baseline FEV1 (< FEV1 50%). SABA reversibility of FEV1 is sufficient to define asthma in absence of MCh PC20.
  4. Subject's asthma has been stable for the past 30 days.
  5. The subject has been a non-smoker for the past year and should have less than a 10 pack year history.
  6. The subject must be capable of and willing to provide written informed consent
  7. The subject is able to understand and comply with protocol requirements and timetables, instructions and protocol-stated restrictions.
* Healthy Subject Inclusion Criteria

  1. Subject is an adult male or female between 18 and 65 years of age inclusive. (Subjects will be age and gender matched) With age matching, we will enroll in a manner that age and gender will be matched 1:1 in the following cohorts: age 21-30, 31-40, 41-50, 51-60, 61-65.
  2. Subject must have an exclusion of asthma or other significant pulmonary diseases (i.e., cystic fibrosis, tuberculosis, Interstitial Lung Disease and bronchopulmonary dysplasia)
  3. The subject has been a non-smoker for the past year and should have less than a 10 pack year history.
  4. The subject has a negative methacholine test (PC20 > 16) and does not use inhaled steroids and/or SABA.
  5. The subject must be capable of and willing to provide written informed consent
  6. The subject is able to understand and comply with protocol requirements and timetables, instructions and protocol-stated restrictions.

     -

     Exclusion Criteria:

  <!-- -->

  1. As a result of the medical interview, physical examination or screening investigations, the physician responsible considers the volunteer unfit for the study.
  2. The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer), prior to the current study.
  3. No oral steroids within the last 3 months.
  4. No current anticoagulant and/or antiplatelet therapy.
  5. The subject has a history of alcohol or drug abuse within the last 5 years.
  6. The subject has history of hepatitis B, hepatitis C, or HIV virus.
  7. The subject has a history of chemotherapy or radiotherapy within the last 2 years.
  8. The subject has a history of diabetes.
  9. The subject is pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 severe asthma subjects matched with 10 healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To obtain bronchial brushings and bronchial alveolar lavage fluid from 10 subjects with severe asthma (GINA criteria in The Global Initiative for Asthma, http://www.ginasthma.org ) and from 10 matched normal healthy subjects. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Reynold Panettieri, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Airways Biology Initiative at the University of Pennsylvania, Philadelphia, Pennsylvania, United States